CLINICAL TRIAL: NCT02522468
Title: A Randomized Single-Center Superiority Trial of Radioactive Seed Localization Versus Needle Localization for Malignant Breast Disease.
Brief Title: A Trial of RSL Versus WL for Malignant Breast Disease
Acronym: BCS-RSL-001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCI-BRE-BCS-RSL-001
Record Dates: First submitted 2015-07-28; First posted 2015-08-13 (Estimated); Last update posted 2022-08-10 (Actual); Status verified 2022-01

CONDITIONS: Breast- Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radioactive Seed Localization (Experimental): Radioactive Seeds
  Interventions: Procedure: Radioactive Seed Localization
- Wire Localization (Active Comparator): Wire
  Interventions: Procedure: Wire Localization

INTERVENTIONS:
Procedure: Radioactive Seed Localization
  Arms: Radioactive Seed Localization
Procedure: Wire Localization
  Arms: Wire Localization

SUMMARY:
The purpose of this randomized trial is to determine the superiority of utilizing radioactive seed localization (RSL) over wire-guided localization (WL) for palpable or non-palpable malignant lesions in patients undergoing breast conservation surgery (BCS).

DETAILED DESCRIPTION:
Consented and eligible subjects will be randomized to either radioactive seed localization or wire localization and stratified by surgeon and invasive versus DCIS prior to localization. Subjects on both arms will undergo breast conservation surgery including surgical specimen removal. Specimens will be grossed according to standard of care procedures. Localization, breast conservation surgery, and post-operative appointments will follow standard of care guidelines. Surveys will be administered according to the study calendar to the radiologist, surgeon, pathologist, and subject for data collection.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 20 to 99 years of age
* Breast lesion necessitating image-guided excision
* Unifocal disease
* Breast-conservation candidate
* Biopsy-proven malignant breast lesion including by not limited to invasive ductal carcinoma, invasive lobular carcinoma, and ductal carcinoma in situ
* Signed written informed consent document by the subject and/or a LAR

Exclusion Criteria:

* Male
* Multifocal or multicentric disease
* Receiving neoadjuvant chemotherapy
* Pregnant or breastfeeding
* Locally advanced disease
* Breast conservation contraindication such as inability to receive whole breast radiation therapy, inability to tolerate localization procedure, inability to lay flat or prone for radiation, and undesirable tumor to breast ratio
* Prior breast cancer on ipsilateral side
* Unable or unwilling to adhere to post-localization instructions (e.g. timely seed removal)

Ages: 20 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2015-07-24 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Surgical Resection Margins | 30 days
  The primary objective for this study will be the comparison between Radioactive Seed Localization (RSL) and Wire-Guided Localization (WL) based on negative margins in malignant breast disease. This is defined as no tumor on ink in invasive disease and greater than or equal to 2mm from the inked margin in non-invasive disease (DCIS).

CONTACTS AND LOCATIONS:
Overall Officials: Lejla Hadzikadic-Gusic, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

DOCUMENTS (1):
  • Informed Consent Form (2015-06-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT02522468/ICF_000.pdf